CLINICAL TRIAL: NCT03082157
Title: Mighty Men Nashville: A Faith-Based Weight Loss Program to Address Cancer Disparities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Transfer of grant to new institution
Sponsor: Vanderbilt University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Derek Griffith, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191252
Record Dates: First submitted 2017-03-10; First posted 2017-03-17 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a community based, cluster randomized, parallel group longitudinal trial. Each faith-based organization that meets inclusion criteria, agrees to participate and sign the memorandum of agreement will be matched on congregation size and randomized to either: 1) the exercise-only comparison group or 2) the Mighty Men weight-loss intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mighty Men Intervention (Experimental): Mighty Men weight-loss intervention including health education and exercise during small group sessions
  Interventions: Behavioral: Mighty Men Intervention
- Comparison (No Intervention): Exercise-only small group sessions

INTERVENTIONS:
Behavioral: Mighty Men Intervention — African American men assigned to this condition will receive: tailored goals/ messages, self-monitoring, small group meetings and educational and community-based information and resources.
  Arms: Mighty Men Intervention

SUMMARY:
Mighty Men is a 6-month faith-based weight-loss intervention for obese African American men 35-74 years old being conducted in Nashville, TN.

DETAILED DESCRIPTION:
Mighty Men is a 6-month faith-based weight-loss intervention for obese African American men 35-74 years old. The investigators will conduct this intervention in African American faith-based organizations because these organizations have the opportunity to consistently reach more African American men than any other institution in the African American community. African American faith-based organizations have historically served as a trusted institution for filling gaps in health and social services, including cancer prevention and control programs, within their natural role and function in the African American community. Additionally, African American faith-based organizations are important resources and sources of information for large numbers of middle-aged and older African American men, including those who are not members of a faith-based organization. Though African American men attend faith-based organization's at lower rates than African American women, men constitute 40% of the congregation membership among the largest denominations serving African Americans.

Mighty Men includes: (a) tailored goals/ messages, (b) self-monitoring, (c) small group training and education and (d) educational and community-based information and resources. There are three specific aims for the proposed study:

Specific Aim 1 is to compare the efficacy of Mighty Men to an attention control group in a cluster-randomized clinical trial of 448 African American men. The investigators hypothesize that men in faith-based organizations assigned to the intervention group will have lost more weight than men in faith-based organizations assigned to the comparison group at 6-months, and they will maintain greater weight loss than men in the control group 3-months post intervention.

Specific Aim 2 is to compare changes in cancer risk behaviors (e.g., healthy eating and physical activity), adiposity measures (e.g., body fat), and psychosocial mediators (e.g., perceived social support, autonomous motivation) at 6-months and 3-months post intervention between Mighty Men and comparison participants. The investigators hypothesize that men assigned to Mighty Men will demonstrate and maintain greater improvements in eating and physical activity and psychosocial mediators than those randomized to the attention control group.

Specific Aim 3 is to examine the impact of Mighty Men on the faith-based organizations that participate in the intervention. The investigators will conduct a rigorous process and impact evaluation to determine the extent of program reach, efficacy, adoption, implementation and maintenance (RE-AIM) in African American faith-based organizations in the intervention condition. Also, investigators hypothesize that faith-based organizations assigned to the intervention will demonstrate greater perceived efficacy to conduct and sustain health ministries for African American men and improvements in all areas of the RE-AIM framework than faith-based organizations randomized to the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* 35-77 at enrollment
* Black/African American
* Male; Less than 400 pounds
* BMI: 27-50
* Fluent in english
* provides informed consent

Exclusion Criteria:

* Pre-existing condition that prohibits at least moderate physical activity
* Serious medical condition that is likely to hinder accurate measurement of weight
* a condition for which weight loss is contraindicated
* a condition that would cause weight loss
* Prior (2 years) or planned (6 months) bariatric surgery
* Chronic use of medications that are likely to cause weight gain or cause weight loss
* No cell phone or land-line phone
* Participant in another obesity, eating or physical activity program or study
* Psychiatric hospitalization or in-patient substance abuse treatment in the past 12 months

Ages: 35 Years to 77 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Most weight loss, healthy eating and physical activity interventions for African Americans have included considerably more African American women than African American men. One of the most crucial challenges in behavioral interventions has been reaching African American men and identifying settings where interventions are sustainable over time. In the past 25 years, no community-based intervention has produced clinically significant changes in weight loss, eating practices or physical activity in African American men. The investigators propose to develop and test the first individually-tailored, weight loss intervention for African American men.
Enrollment: 0 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 6 months post-baseline
  The Primary outcome is change in weight loss at 6-months post-baseline.

SECONDARY OUTCOMES:
Dietary patterns | 6 months post-baseline
  Dietary patterns will be assessed using tools to measure fruit and vegetable intake and fat intake. Fruit and vegetable intake will be assessed using servings of fruits and vegetables consumed per day assessed with two brief frequency measures.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Griffith, PhD, Principal Investigator — Vanderbilt University; Emily C Jaeger, MPH, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffith DM, Pennings JS, Jaeger EC. Mighty Men: A Pilot Test of the Feasibility and Acceptability of a Faith-Based, Individually Tailored, Cluster-Randomized Weight Loss Trial for Middle-Aged and Older African American Men. Am J Mens Health. 2023 Jul-Aug;17(4):15579883231193235. doi: 10.1177/15579883231193235. PMID 37608590
- See also: Mighty Men: A faith-based weight loss intervention to reduce cancer risk in African American men — https://books.google.com/books?hl=en&lr=&id=zHzZDwAAQBAJ&oi=fnd&pg=PA189&dq=Mighty+Men:+A+Faith-based+Weight+Loss+Intervention+to+Reduce+Cancer+Risk+in+African+American+Men&ots=8TD3aUOpxz&sig=9_hjRbAfu_PEMUgw_tGvKJCYN50#v=onepage&q=Mighty%20Men%3A%20A%20Faith-based%20Weight%20Loss%20Intervention%20to%20Reduce%20Cancer%20Risk%20in%20African%20American%20Men&f=false